CLINICAL TRIAL: NCT06600100
Title: Inhibitory Control Training for the Treatment of Excess Weight: Behavioural, Cognitive and Anthropometric Changes (InhibeT)
Brief Title: Inhibitory Control Training for Excess Weight: Behavioural, Cognitive and Anthropometric Changes
Acronym: InhibeT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raquel Vilar López (Other)
Collaborators: Government of Spain (Unknown)
Responsible Party: Sponsor-Investigator, Raquel Vilar López, Principal Investigator, Universidad de Granada
Organization: Universidad de Granada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID2022-137524OB-I00
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity; Inhibition, Psychological
Keywords: excess weight; overweight; inhibitory control training; FoodT
MeSH Terms: conditions — Overweight; Obesity; Inhibition, Psychological | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitory control training (Experimental): Inhibitory control training using the active version of the FoodT App. An experimental group will receive: i) an informative session; ii) 3 pre-treatment sessions (one assessment with questionnaires and two counselling sessions: one on diet and one on physical exercise); iii) A psychology session in which the investigator will explain the task to participants and the procedure for the next two weeks. A daily reminder will be sent by WhatsApp to the participants' phone to train for 10 minutes a day from Monday to Friday for two weeks; iv) a session of post treatment assessment (questionnaires); v) one follow-up session three months after completing the intervention to repeat the evaluation
  Interventions: Behavioral: Inhibitory control training
- Placebo inhibitory control training (Placebo Comparator): Placebo inhibitory control training using the placebo version of the FoodT App. The placebo group will receive: i) an informative session; ii) 3 pre-treatment sessions (one assessment with questionnaires and two counselling sessions: one on diet and one on physical exercise); iii) A psychology session in which the investigator will explain the task to participants and the procedure for the next two weeks. It won't be necessary to meet every day; A daily reminder will be sent by WhatsApp to the participants' phone to train for 10 minutes a day from Monday to Friday for two weeks; iv) a session of post treatment assessment (questionnaires); v) one follow-up session three months after completing the intervention to repeat the evaluation
  Interventions: Behavioral: Placebo Inhibitory control training

INTERVENTIONS:
Behavioral: Inhibitory control training — Computerized cognitive training. Participants will perform the task of the FoodT app for 10 minutes during two weeks (taking advantage of time of maximum brain potentiation, Rossi et al., 2009). Images of food and non-food appear on the left, right or centre of the smart phone screen and participants must touch it (or not, depending on the cue) with their index finger as quickly as possible. Participants earn points for correct tap responses and lose points for incorrect tap responses. If the image has a green border around it, participants must tap the image and win 1 point. But if the image has a red border around it, participants must inhibit the tapping response, or lose 1 point. Participants must respond as quickly and accurately as possible. Pictures of healthy and unhealthy foods are always paired with the Go and the No-Go signal, respectively. Non-food images are paired 50% of the time with the Go and the No-Go signal
  Other Names: FoodT (active)
  Arms: Inhibitory control training
Behavioral: Placebo Inhibitory control training — Computerized cognitive training. Participants will perform the task of the FoodT app for 10 minutes during two weeks (taking advantage of time of maximum brain potentiation, Rossi et al., 2009). Images appear on the left, right or centre of the smart phone screen and participants must touch it (or not, depending on the cue) with their index finger as quickly as possible. Participants earn points for correct tap responses and lose points for incorrect tap responses. If the image has a green border around it, participants must tap the image and win 1 point. But if the image has a red border around it, participants must inhibit the tapping response, or lose 1 point. Participants must respond as quickly and accurately as possible. Here, three separate categories of non-food items (stationery, flowers and clothing) would be Go signal (associated with green 100%), No-Go signal (associated with red 100%) and control (50% red 50% green) respectively.
  Other Names: FoodT (placebo)
  Arms: Placebo inhibitory control training

SUMMARY:
People with excess weight (EW) are characterized by high impulsivity, high levels of craving for high-calorie foods, deficits in inhibitory control, and maladaptive decision-making. The proposed intervention seeks to target these issues. Thus, the present study aims to determine the effectiveness of combining inhibitory control training with usual treatment (diet and physical exercise) in treating people with EW to produce cognitive, behavioral and anthropometric changes. Participants will be randomly allocated to one of two groups: 1) the experimental group that would receive active inhibitory control training and (2) the active control group that will receive placebo inhibitory control training. Both groups will receive individualized diet and physical exercise guidelines. Training requires to inhibit responding to certain foods presented during computerized tasks. Using a food Go/No-Go paradigm, individuals are asked to press a button when a Go cue is presented next to an image and to refrain from pressing a button when a No-Go cue (e.g., a bold frame) is presented. In the experimental group, pictures of healthy and unhealthy foods are always paired with the Go and the No-Go signal, respectively whereas in the control group healthy and unhealthy foods are paired 50% of the time with the Go and 50% with the No-Go signal. It is hypothesized that the experimental intervention would be effective improving (i) Body Mass Index (BMI), (ii) food craving, (iii) anthropometric measures (waist circumference and waist-to-hip and waist-to-height ratios), (iv) eating and physical exercise behaviors (decreased caloric intake and increased frequency and time of physical activity), (v) emotional symptoms and emotional eating (depression, anxiety, emotional regulation, emotional eating, reward-related eating, non-homeostatic eating), and (vi) cognitive abilities (motor and cognitive inhibition, delay of gratification, impulsivity, working memory, cognitive flexibility and decision making).

DETAILED DESCRIPTION:
1. HYPOTHESIS: Inhibitory control training with the food Go/NoGo paradigm will be effective in treating people with EW. Thus, the active intervention, compared to the placebo, will achieve: (i) decreased BMI, (ii) decreased craving, (iii) improved anthropometric measures (waist circumference and waist-to-hip and waist-to-height ratios), (iv) improved eating and exercise behaviors (decreased caloric intake increased frequency and time of physical activity), (v) improved emotional symptoms and emotional eating (depression, anxiety, emotional regulation, emotional eating, reward-related eating, non-homeostatic eating), (vi) improved cognitive abilities (motor and cognitive inhibition, delay of gratification, impulsivity, working memory, cognitive flexibility and decision making).

   GENERAL OBJECTIVE: To determine the effectiveness of inhibitory control training for the treatment of people with EW (improvements in BMI, craving, anthropometric measures, food and physical exercise behaviours, emotional symptoms and emotional eating, and cognitive measures).
2. METHODOLOGY

   2.1. Design: Randomized controlled trial of parallel groups. The sample size calculation was performed with the G*Power 3.1 tool. To do so, it will be relied on the only study to date that applied food Go/NoGo training (4 sessions in one week) on a median effect size for reducing BMI post-treatment (Cohen's d = 0.57) and at 6-month follow-up (Cohen's d = 0.48). Thus, considering a median effect size for conducting ANOVAs (f= 0.25), the minimum recommended N to reach a power of 0.80, assuming an alpha level of 0.05 with two groups and three repeated measures, was 44 participants, 22 per group. Nevertheless, a conservative approach will be adopted and decided to increase groups to 27 participants.

   The participants (N=54) will be randomly allocated to two groups: (i) experimental group (active inhibitory control training); n=27 and (ii) active control group (placebo inhibitory control training); n=27).

   2.3. Interventions

   Pre-treatment sessions: information, dietary plus physical guidelines (all groups):

   First, all participants will participate in a group briefing informational session about the procedure and rationale of the study that will last about an hour. Also, informative videos and brochures will be provided. There will be two 90-minute sessions afterwards given by a nutritionist and personal trainer respectively to provide individualized diet and physical exercise instructions to all participants.

   Cognitive interventions (both groups): Duration: 2 weeks in which participants should train from monday to friday for 10 minutes with the active or the placebo version of the Food Trainer App (FoodT) with their smart phones.

   2.4. Outcome measures: change in Body Mass Index (BMI) will be the main outcome measure. Secondary outcomes will be changes in food craving, anthropometric measures, eating and physical activity behaviours, emotional symptoms and emotional eating, and cognitive measures. Screening and descriptive measured will include a sociodemographic questionnaire, depression and anxiety questionnaires, motivation and questionnaire on Eating and Weight Patterns-5.
3. PROCEDURE The whole study will be delivered online. Inclusion and exclusion criteria will be checked through the data collected in a questionnaire of sociodemographic and clinical variables. Further, psychopathology exclusion criteria will be tested with three questionnaires to measure depression, anxiety, and stress symptoms as well as binge eating and bulimia (BDI, DASS-21 and QEWP-5), and a short clinical interview by phone and/or information requested by email in those cases where there are doubts about any of the aspects collected through the online instruments.

All candidates who meet the criteria will attend an information meeting about the project in which participants will receive written and oral information and will be asked for their informed consent. Then, participants will be randomly assigned to groups before the pre-treatment assessment sessions. Both groups of the study (experimental and active control) will complete pre and post assessments, as well as the 3-month follow-up (see below). What will differentiate the groups will be, therefore, the treatment: active vs. placebo inhibitory control training. If at the end of the project the active training has proven to be effective, the control group will be offered the possibility to carry out the active training.

All sessions will be developed in groups of 4-6 people. There will be at least 5 groups of intervention sessions (27 participants) and 5 groups for the placebo condition (27 participants). The program will comprise 6 weeks including three assessments (pre, post and 3-month follow-up), two FoodT training weeks, as well as the information and nutrition and exercise sessions. Assessment sessions will last about 2 hours each while the inhibitory control training will last 10 minutes per day.

1. Informative session (session 1; week 1): For the participants to understand the foundation of the intervention information about the aims, basis of the project and the procedure of the research will be given. Participants will be provided written informed consent as well. At the end of this session, participants will be asked for their informed written consent.
2. Pre-treatment assessment (session 2; week 2): All participants will complete the following instruments to assess the main and secondary outcomes, and the exploratory and economic measures: WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, FCQ-S-r, CFA, IPAQ, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36, SOCRATES 00, QEWP-5, sociodemographic questionnaire, another one about used health resources, stigma and previous treatments questions.
3. Nutrition and exercise sessions (session 3; week 3): Participants will receive information on healthy nutritional (Ph.D. Nutritionist) and physical exercise (Ph.D. Sports Science professional) habits. In addition, participants will receive individualized diet and physical exercise guidelines, and participants will be able to consult any doubts to both professionals through WhatsApp groups.
4. Training sessions (sessions 4 to 14, weeks 4 and 5): A daily reminder will be sent by WhatsApp to the participants' phone to train from Monday to Friday during 10 minutes for two weeks. The FoodT app will be used to pair high-calorie meals with the no-go cue. Images can appear on the left, right or center of the screen, and should be tapped or not depending on whether the image has a green or red circle around them. Participants earn points for correct tapping responses and lose points for incorrect tapping responses and must respond as quickly and accurately as possible. The placebo FoodT has images of objects rather than food.
5. Post-treatment assessment (session 15; week 6): To evaluate the effectiveness of the interventions, BMI and the following instruments will be administered to obtain the main and secondary outcomes: FCQ-T/S-r, WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, CFA, IPAQ, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36, and a questionnaire about used health resources.
6. Follow-up (session 16; week 18): Follow-up at 3 months after the intervention will include the following measures: FCQ-T/S-r, WCST, Food Go/NoGo, IGT, Stroop, Food DD, N-Back, FCQ-S-r, CFA, IPAQ, DASS-21, BDI-II, PEMS, RED, DEBQ, PSRSQ, ERQ, UPPS-P, SF-36 and a questionnaire about used health resources. Anthropometric measures will be repeated as well. Every month after the end of the treatment, participants will be contacted by email and mobile message to maintain adherence.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 39.9
* Age between 18 and 60 years
* Proficiency in the Spanish language
* Internet access
* Computer and smartphone

Exclusion Criteria:

* Traumatic, digestive, metabolic or systemic disorders that affect the central nervous system, autonomic or endocrine
* Severe psychopathological disorders, moderate depressive symptoms or treatment for depression
* Eating disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI). Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  BMI is a measure of body fat based on height and weight. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m^2. Height and weight will be obtained with a pharmacy digital weight.

SECONDARY OUTCOMES:
Food Craving. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Change in food Craving. Food Craving Questionnaire State-reduced (FCQ-S-r)consists of 15 items to be scored on a 5-point scale ranging from strongly disagree to strongly agree. A higher score indicates higher state of craving at the time of the assessment
Waist circumference (WC). Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)]
  To take these measurements at home, participants should ask someone for help and follow our instructions. WC will be measured in cm with a tape around the waist, just above the navel.
Waist-to-hip ratio (WHR). Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)]
  To take these measurements at home, participants should ask someone for help and follow our instructions. WHR results from WC divided by the hip circumference in cm (tape placed at the maximum prominence of the buttocks).
Waist-to-height ratio (WHtR). Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)]
  To take these measurements at home, participants should ask someone for help and follow our instructions. WHtR results from WC divided by the height measured standing with heels close together and trunk erect.
Eating behaviour. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)]
  Diet information during the last year (pre-treatment), two last weeks (post-treatment) and 3 last months (follow-up) will be collected through a 52-item Food frequency questionnaire (CFA). Participants must record quantities of all the foods and drinks consumed during those periods. Data are transformed into total calories and calories from fats, carbohydrates, and sugars
Physical activity behaviour. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)]
  International Physical Activity Questionnaire (IPAQ; www.ipaq.ki.se): is a questionnaire with 7 questions on physical activity during the last week, as well as walking and sitting time.It evaluates physical activity related to work, activity at home and free time determines the degrees of activity based on the metabolic equivalents (MET) consumed.Higher scores indicate greater physical activity
Anxiety and Stress. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Depression Anxiety Stress Scale-21 (DASS-21) will be used, taking into account scores on the stress and anxiety subscales. The scores for both subscales range from 0 to 21, a higher score indicating higher anxiety or stress.
Depression symptoms. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Beck Depression Inventory will be administered to test depression symptoms.The scores range from 0 to 63 points. The higher the score, the greater the severity of depressive symptoms.
Non homeostatic eating. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Dutch Eating Behaviour Questionnaire (DEBQ) will be administered to assess restrictive eating behaviours related to external cues and emotional states. Higher scores in each subscale reflect higher level of restrained, emotional, and external eating, respectively.The DEBQ uses a 5-point Likert scale, ranging from never (1) to very often (5). The average score is calculated for each subscale by adding scores obtained from individual items and dividing them by the number of items included in a subscale (mean range: 1-5).
Reward-related eating. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Reward-Based Eating Scale (RED) is a 13 items questionnaire that evaluates worries about foods, losing intake control and absence of satiety. Higher scores reflect higher reward-based eating drive.
Emotional eating. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Coping subscale of the Palatable Eating Motives Scale (PEMS) will be used to evaluate the intentionality for eating palatable foods to face negative emotions. The coping subscale includes items that are scored on a 5-point Likert-type scale, the total range being from 5 to 25 points. Low scores indicate that the person rarely resorts to the consumption of pleasant foods as a strategy to cope with negative emotions or stressful situations. High scores suggest that the person frequently uses palatable food as a strategy to cope with stress or negative emotions, which may be related to unhealthy eating habits or emotional eating patterns.
Emotion Regulation Strategies. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  The Emotion Questionnaire (ERQ) consists of 10 items to examine cognitive reappraisal and expressive suppression strategies. In cognitive reappraisal the highest score (42) is associated with better emotional outcomes while in expressive suppression the highest score (28) is linked to poorer well-being. Each item is rated on a Likert scale from strongly disagree (1) to strongly agree (7).
Motor inhibition. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Motor inhibition will be assessed using FoodT. In the FoodT app reaction time for the high-calorie and low-calorie foods paired with the go and the no-go signal. The average response time for go and no-go items will be calculated according to the type of images (appetizing and healthy foods), and commission errors will be recorded.
Cognitive inhibition. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Using a Stroop task with food, the interference of food-related words on task performance can be measured as an assessment of cognitive inhibition.
Delay of gratification. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Score on the Food Delay Discounting will be used to measure the sensitivity to immediate rewards vs higher value rewards delayed. The participant's choices are recorded for each trial. Each trial varies in terms of the amount of reward and the amount of time to wait. To model the decisions, a hyperbolic discounting function is generally used.
Inhibition and activation systems. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  This will be assessed using the Punishment Sensitivity and Reward Sensitivity Questionnaire (PSRSQ) of 48 items. Responses in the scale are in a "yes/no" format. Higher punishment sensitivity scores are associated with lower number of punishable errors while higher reward sensitivity punctuations are linked to higher number of passive avoidance errors.
Self-reported impulsivity. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Self-reported impulsivity will be measured with Impulsive behaviour scale (UPPS-P). It consists of 20 items scored on a four point Likert scale, ranging from strongly agree (1) to strongly disagree (4). Higher scores mean worse outcome in impulsivity, while lower scores are related to better self-control and regulation
Working Memory. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Working Memory will be assessed using N-back Task score based on accuracy and reaction times. Higher accuracy scores indicate stronger working memory and attention, while faster reaction times are linked to quicker processing speed and decision-making.
Cognitive flexibility. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Wisconsin Card Sorting Test will be administered to measure shift strategy in response to changing contingencies. There are128 trials where more correct responses, fewer perseverative and non perseverative errors, and more completed categories (max 6) are related to better performance.
Decision making. Mean change from baseline at post-intervention | Pre-treatment assessment (week 2), post-treatment assessment (week 6) and follow-up (week 18)
  Iowa Gambling Task will be used to assess decision-making using money rewards.

OTHER OUTCOMES:
Descriptive measures | Pre-treatment assessment (week 2)
  A socio-demographic questionnaire will be administered to examine age, education, gender, socio-economic variables and clinical variables to consider exclusion and inclusion criteria. All these variables are qualitative.
Depression Symptoms . Screening | Pre-treatment assessment (week 2)
  The Beck Depression Inventory (BDI-II) will also be used to rule out major depressive symptoms as an exclusion criteria. The scores range from 0 to 63 points. Participants with a score higher than 29, indicative of severe symptoms, will be excluded.
Anxiety Symptoms . Screening | Pre-treatment assessment (week 2)
  The anxiety subscale of the DASS-21 will also be used to rule out symptoms of major anxiety as an exclusion criterion. The scores for both subscales range from 0 to 21. Participants with a score higher than 8, indicative of severe symptoms, will be excluded from the study.
Eating and Weight Patterns. Screening | Pre-treatment assessment (week 2)
  Questionnaire on Eating and Weight Patterns-5 (QEWP-5) is adapted to DSM-5 criteria and will be used to exclude people with binge eating problems and bulimia. The QEWP-5 is not scored on a traditional numerical scale like other psychological tests; instead, responses are used to identify the presence of eating disorder symptoms. Positive responses to key questions about the frequency of binge eating, compensatory behaviors, and emotional distress may indicate the presence of an eating disorder.
Using of Health Resources. | Pre-treatment assessment (week 2)
  The Health Resources Questionnaire asks how often and why people have needed medical care and medicines in the last 3 month to measure the impact of the intervention in terms of health uses. Fewer visits to health professionals will be indicative of improvement.
Motivation to change. | Pre-treatment assessment (week 2)
  Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) adapted to excess weight will be used to assess motivation to change habits. It has 18 items that score readiness to change in people with abusive food use with a five point Likert scale, ranging from strongly disagree (1) to strongly agree (5). Higher scores mean better outcome in relation to motivation to change, while higher scores on ambivalence suggest doubts about the motivation to change.
Stigma. | Pre-treatment assessment (week 2)
  A yes/no question will be asked to record whether or not participants have experienced weight stigma in the past.
Previous treatment history | Pre-treatment assessment (week 2)
  History of previous treatment, from pharmacological or nutritional to psychological, should be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vilar López, Ph.D, Principal Investigator — Universidad de Granada
Locations (1):
- Mind, Brain and Behavior Research Center at University of Granada (CIMCYC), Granada, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee and who provide a methodologically sound proposal. Proposals should be directed to rvilar@ugr.es

REFERENCES:
- See also: Project website — http://trainep.ugr.es/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT06600100/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT06600100/ICF_003.pdf